CLINICAL TRIAL: NCT00476021
Title: Randomized Trial of Postplacental or Delayed Insertion of the Levonorgestrel-releasing Intrauterine Device After Vaginal Delivery
Brief Title: Postplacental or Delayed Insertion of the Levonorgestrel-releasing Intrauterine Device (IUD) After Vaginal Delivery
Acronym: POPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Beatrice Chen, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO06070007
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Contraception
Keywords: postpartum; contraception; postplacental IUD; intrauterine devices

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postplacental IUD insertion (Experimental): immediate postplacental levonorgestrel-releasing IUD (Mirena) insertion
  Interventions: Device: Levonorgestrel-releasing IUD (Mirena)
- Delayed IUD insertion (Active Comparator): delayed levonorgestrel-releasing IUD (Mirena) insertion (6-8 weeks after delivery)
  Interventions: Device: Levonorgestrel-releasing IUD (Mirena)

INTERVENTIONS:
Device: Levonorgestrel-releasing IUD (Mirena) — levonorgestrel-releasing IUD containing 52 mg levonorgestrel, indicated for use for up to 5 years
  Other Names: Mirena

SUMMARY:
This study is a randomized controlled trial comparing 6 month usage rates of the levonorgestrel-releasing intrauterine device (LNG-IUD) when inserted postplacentally after vaginal delivery or delayed placement at 6-8 weeks postpartum. Given the high rate of unintended pregnancy in the United States, particularly in postpartum women, there is a need for reliable, effective, long-term contraception such as the IUD in postpartum women. Postplacental insertion of intrauterine contraception would help to address this need. The primary hypothesis of this study is that use of the LNG-IUD at 6 months after vaginal delivery will be higher in women who have immediate postplacental insertion as compared to delayed insertion 6-8 weeks following delivery.

DETAILED DESCRIPTION:
The United States (US) has the highest unintended pregnancy rate of any developed country. Of the 6.4 million pregnancies in the US each year, almost half are unintended (49%). Roughly half of these (22% of all pregnancies) result in unintended births, while 20% of all pregnancies result in abortion. Postpartum women are particularly susceptible, with an unintended pregnancy rate of 10%-44% in the first year postpartum. These unintended pregnancies occur despite the recommendation that a contraceptive method be selected prior to hospital discharge.

Given the high rate of unintended pregnancy in the United States, particularly in postpartum women, there is a need for reliable, effective, long-term contraception such as the IUD in postpartum women. Postplacental insertion of intrauterine contraception would help to address this need. The IUD is a highly effective but underused method of postpartum contraception. Although the expulsion rate in postplacental insertion is higher than interval insertion, the benefits of highly effective contraception available immediately after delivery may outweigh the risks of expulsion.

To date, there have been no randomized trials of postplacental insertion of the LNG-IUD in the United States. One pilot study in the United States of 20 subjects who received an ultrasound-guided postplacental insertion of the LNG-IUD showed an acceptable expulsion rate of 10% and no infections over a 10-week follow-up, thus making postplacental insertion of LNG-IUD safe for further study.

This study is a randomized controlled trial comparing 6 month usage rates of the levonorgestrel-releasing intrauterine device (LNG-IUD) when inserted postplacentally after vaginal delivery or delayed placement at 6-8 weeks postpartum. One hundred sixty-eight women receiving prenatal care at Magee-Womens Hospital, Pittsburgh, PA, who are interested in using the LNG-IUD for contraception will be enrolled during their pregnancy. The IUD will be inserted within 10 minutes after delivery of the placenta in women randomized to immediate insertion. Delayed IUD insertion will be performed at the first postpartum visit in 6-8 weeks. All subjects will follow up in person at 6-8 weeks and 6 months after delivery. A telephone interview will occur at 3 months after delivery for all subjects.

Subjects who are not eligible for insertion due to post-randomization ineligibility criteria will be referred to their primary gynecologist or midwife for delayed IUD placement. They will be contacted by phone at 3 and 6 months to assess quality of life, contraceptive usage, and unintended pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Greater than or equal to 24 0/7 weeks pregnant at time of enrollment
* Anticipates undergoing a vaginal delivery
* Desires to use the LNG-IUD (Mirena) for postpartum contraception
* Willing and able to sign an informed consent in English
* Willing to comply with the study protocol

Exclusion Criteria:

* Planning to undergo a scheduled cesarean section
* Allergy to either polyethylene or levonorgestrel or other contraindications to use of the LNG-IUD
* Exposure to or treatment for gonorrhea, chlamydia, or trichomoniasis during the pregnancy
* Presence of one or more leiomyomata greater than 3 centimeters in diameter
* Uterine anomaly (other than a repaired septate uterus)
* Current cervical cancer or carcinoma in-situ
* Desires repeat pregnancy within one year of delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice A Chen, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chen BA, Reeves MF, Hayes JL, Hohmann HL, Perriera LK, Creinin MD. Postplacental or delayed insertion of the levonorgestrel intrauterine device after vaginal delivery: a randomized controlled trial. Obstet Gynecol. 2010 Nov;116(5):1079-87. doi: 10.1097/AOG.0b013e3181f73fac. PMID 20966692
- [Result] Chen BA, Reeves MF, Creinin MD, Schwarz EB. Postplacental or delayed levonorgestrel intrauterine device insertion and breast-feeding duration. Contraception. 2011 Nov;84(5):499-504. doi: 10.1016/j.contraception.2011.01.022. Epub 2011 Apr 16. PMID 22018124
- See also: Click here for more information about the Center for Family Planning Research, University of Pittsburgh — http://www.birthcontrolstudies.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Postplacental IUD Insertion: Postplacental LNG-IUD insertion
- Delayed IUD Insertion: Delayed LNG-IUD insertion
Period: Overall Study
Arm/Group | Postplacental IUD Insertion | Delayed IUD Insertion
Started | 51 | 51
Completed | 51 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Immediate Postplacental IUD Insertion: immediate postplacental IUD insertion
  Levonorgestrel-releasing IUD (Mirena): levonorgestrel-releasing IUD containing 52 mg levonorgestrel, indicated for use for up to 5 years
- Delayed IUD Insertion (6-8 Weeks After Delivery): delayed IUD insertion (6-8 weeks after delivery)
  Levonorgestrel-releasing IUD (Mirena): levonorgestrel-releasing IUD containing 52 mg levonorgestrel, indicated for use for up to 5 years
- Total: Total of all reporting groups
Arm/Group | Immediate Postplacental IUD Insertion | Delayed IUD Insertion (6-8 Weeks After Delivery) | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 51 | 102
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (5.3) | 24.7 (5.2) | 25.1 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 102
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 51 | 102
Received IUD per protocol [Number; unit: participants]
  Received IUD per protocol | 50 | 46 | 96
  Did not receive IUD per protocol | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: IUD Usage Rate at 6 Months
Description: Usage rate of the LNG-IUD at 6 months after delivery
Time Frame: 6 months after delivery
Population: IUD use at 6 months, lost to follow-up counted as failures
Measure: Number; unit: participants
Arm/Group | Postplacental IUD Insertion | Delayed IUD Insertion
Number analyzed (Participants) | 51 | 51
participants | 43 | 39

2. Secondary Outcome: Proportion of Women Who Are Able to Have the LNG-IUD Placed Postplacentally and Are Not Excluded From Placement
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Received Postplacental IUD: Received postplacental LNG-IUD
Arm/Group | Received Postplacental IUD
Number analyzed (Participants) | 51
participants | 50

3. Secondary Outcome: Follow-up Rates for Delayed Insertion of LNG-IUD
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Delayed IUD Insertion: Followed up for delayed IUD insertion
Arm/Group | Delayed IUD Insertion
Number analyzed (Participants) | 51
participants | 46

4. Secondary Outcome: Expulsion Rates of Post-placental and Delayed Insertion of the LNG-IUD Using Clinical Exam and Ultrasonography
Time Frame: 6 months
Population: The population only includes women who received IUDs at the specified timepoint. Only 50/51 women in the postplacental group had a successful IUD insertion postplacentally. Only 46 of 51 women in the delayed group returned for a delayed IUD insertion.
Measure: Number; unit: participants
Arm/Group | Postplacental IUD Insertion | Delayed IUD Insertion
Number analyzed (Participants) | 50 | 46
participants | 12 | 2

5. Secondary Outcome: Safety of Postplacental Insertion of the LNG-IUD as Measured by Infection Rates
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Postplacental IUD Insertion: Infection after postplacental LNG-IUD insertion
- Delayed IUD Insertion: Infection after delayed LNG-IUD insertion
Arm/Group | Postplacental IUD Insertion | Delayed IUD Insertion
Number analyzed (Participants) | 51 | 51
participants | 1 | 1

6. Secondary Outcome: Rates of Follow-up and Unintended Pregnancy Rates for Subjects Who Are Excluded From Postpartum Insertion
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Pregnancy Within 6 Months for Ineligible Participants: If a participant was found to be ineligible as a result of postenrollment criteria, she was instructed to follow up with her primary obstetrician or midwife for postpartum contraception and delayed IUD insertion
- Follow-up for IUD Insertion for Ineligible Participants: Ineligible participants were followed for 6 months to evaluate whether they received an IUD from their ob/gyn
Arm/Group | Pregnancy Within 6 Months for Ineligible Participants | Follow-up for IUD Insertion for Ineligible Participants
Number analyzed (Participants) | 41 | 41
participants | 2 | 11

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Postplacental IUD Insertion | Delayed IUD Insertion
Serious Adverse Events (participants affected / at risk) | 1/51 | 0/51
Other Adverse Events (participants affected / at risk) | 3/51 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Postplacental IUD Insertion (N=51) | Delayed IUD Insertion (N=51)
death (Social circumstances) | 1 (1) | 0 (0) — One participant died as a result of unrelated causes
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Postplacental IUD Insertion (N=51) | Delayed IUD Insertion (N=51)
vaginal laceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) — a participant who underwent a postplacental insertion experienced a vaginal laceration when the IUD strings were cut with scissors, requiring repair with suture
retained IUD insertion tube (Reproductive system and breast disorders) | 1 (1) | 0 (0) — IUD insertion tube appeared to have detached from the IUD inserter and had been left inside her uterus during the postplacental IUD placement. Tihs was considered a complete expulsion for the analysis
malpositioned IUD (Reproductive system and breast disorders) | 1 (1) | 0 (0) — IUD was positioned obliquely in the uterus with the arms of the IUD against the right uterine wall and the base of the IUD in the left cornua. Participant was asymptomatic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes